CLINICAL TRIAL: NCT02267850
Title: Effect of Intra-Oral Photobiomodulation on Orthodontic Treatment Time: A Randomized Control Trial
Brief Title: Effect of Intra-Oral Photobiomodulation on Orthodontic Treatment Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biolux Research Holdings, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TS2
Record Dates: First submitted 2014-10-10; First posted 2014-10-20 (Estimated); Results first posted 2018-03-27 (Actual); Last update posted 2018-09-21 (Actual); Status verified 2018-02

CONDITIONS: Malocclusion
Keywords: Photobiomodulation; Orthodontic treatment; Malocclusion; OrthoPulse™
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- OrthoPulse™ (Experimental): Subjects assigned to this group receive fixed orthodontic appliance treatment in conjunction with receiving daily OrthoPulse™ treatments.
  Interventions: Other: Fixed Orthodontic Appliance Treatment; Device: OrthoPulse™
- Sham-Control OrthoPulse™ (Sham Comparator): Subjects assigned to this group receive fixed orthodontic appliance treatment in conjunction with carrying out daily non-functional OrthoPulse™ treatments (untreated control).
  Interventions: Other: Fixed Orthodontic Appliance Treatment; Device: Non-Functional OrthoPulse™

INTERVENTIONS:
Other: Fixed Orthodontic Appliance Treatment — Patients are treated for full mouth fixed orthodontic appliance treatment by the qualified Principal Investigator (PI). Treatment and follow-up appointments per the traditional practices of the PI and dental office.
Device: OrthoPulse™ — Patients carry out daily OrthoPulse™ treatments at home.
  Arms: OrthoPulse™
Device: Non-Functional OrthoPulse™ — Patients carry out daily sham-OrthoPulse™ treatments at home. This is a non-functional device so patients do not receive photobiomodulation therapy.
  Arms: Sham-Control OrthoPulse™

SUMMARY:
The aim of this study is to determine the effect of OrthoPulse™, an intra-oral LED (Light Emitting Diode) photobiomodulation device, on orthodontic treatment time. This is a double-blinded RCT with half the patients receiving treatment from a sham non-functional device, serving as controls, and the other half receiving light therapy treatment from a functional OrthoPulse™. Orthodontic treatment time for the sham-control patients are compared to that of the OrthoPulse™ patients.

ELIGIBILITY:
Inclusion Criteria:

* Presence of permanent dentition
* Eligible and scheduled for full mouth fixed orthodontic treatment.
* Class I or Class II malocclusion (no more than ½ cusp in Class II)
* Non-extraction in all quadrants
* Non-smoker, non-use of chewing tobacco
* Good oral hygiene
* No adjunct treatment such as extra or intraoral appliances
* Age 12-40

Exclusion Criteria:

* Pregnant females
* Patient is currently enrolled in another clinical study
* Non-steroidal Anti-Inflammatory drug (NSAID) use during study (Acetominophen acceptable)
* Periodontally involved teeth
* Use of bisphosphonates
* Unerupted erupted teeth
* Teeth blocked out of alignment and unable to engage initial arch wire

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 29 (Actual)
Dates: Start 2013-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Shaughnessy, DDS, Principal Investigator — Shaughnessy Orthodontics
Locations (1):
- Shaughnessy Orthodontics, Suwanee, Georgia, United States

REFERENCES:
- [Background] Nimeri G, Kau CH, Corona R, Shelly J. The effect of photobiomodulation on root resorption during orthodontic treatment. Clin Cosmet Investig Dent. 2014 Jan 15;6:1-8. doi: 10.2147/CCIDE.S49489. eCollection 2014. PMID 24470774
- [Background] Ekizer A, Uysal T, Guray E, Akkus D. Effect of LED-mediated-photobiomodulation therapy on orthodontic tooth movement and root resorption in rats. Lasers Med Sci. 2015 Feb;30(2):779-85. doi: 10.1007/s10103-013-1405-3. Epub 2013 Aug 29. PMID 23990217
- [Background] Ekizer A, Uysal T, Guray E, Yuksel Y. Light-emitting diode photobiomodulation: effect on bone formation in orthopedically expanded suture in rats--early bone changes. Lasers Med Sci. 2013 Sep;28(5):1263-70. doi: 10.1007/s10103-012-1214-0. Epub 2012 Nov 9. PMID 23139069
- [Background] El-Bialy T, Alhadlaq A, Felemban N, Yeung J, Ebrahim A, Hassan AH. The effect of light-emitting diode and laser on mandibular growth in rats. Angle Orthod. 2015 Mar;85(2):233-8. doi: 10.2319/030914-170.1. Epub 2014 Jul 14. PMID 25017014
- [Background] Uysal T, Ekizer A, Akcay H, Etoz O, Guray E. Resonance frequency analysis of orthodontic miniscrews subjected to light-emitting diode photobiomodulation therapy. Eur J Orthod. 2012 Feb;34(1):44-51. doi: 10.1093/ejo/cjq166. Epub 2010 Dec 27. PMID 21187526
- [Background] Kau CH, Kantarci A, Shaughnessy T, Vachiramon A, Santiwong P, de la Fuente A, Skrenes D, Ma D, Brawn P. Photobiomodulation accelerates orthodontic alignment in the early phase of treatment. Prog Orthod. 2013 Sep 19;14:30. doi: 10.1186/2196-1042-14-30. PMID 24326198
- [Background] Dias FJ, Issa JP, Vicentini FT, Fonseca MJ, Leao JC, Siessere S, Regalo SC, Iyomasa MM. Effects of low-level laser therapy on the oxidative metabolism and matrix proteins in the rat masseter muscle. Photomed Laser Surg. 2011 Oct;29(10):677-84. doi: 10.1089/pho.2010.2879. Epub 2011 Jul 11. PMID 21745137
- [Background] Silveira PC, Silva LA, Fraga DB, Freitas TP, Streck EL, Pinho R. Evaluation of mitochondrial respiratory chain activity in muscle healing by low-level laser therapy. J Photochem Photobiol B. 2009 May 4;95(2):89-92. doi: 10.1016/j.jphotobiol.2009.01.004. Epub 2009 Jan 21. PMID 19232497
- [Background] Cruz DR, Kohara EK, Ribeiro MS, Wetter NU. Effects of low-intensity laser therapy on the orthodontic movement velocity of human teeth: a preliminary study. Lasers Surg Med. 2004;35(2):117-20. doi: 10.1002/lsm.20076. PMID 15334614
- [Background] Esper MA, Nicolau RA, Arisawa EA. The effect of two phototherapy protocols on pain control in orthodontic procedure--a preliminary clinical study. Lasers Med Sci. 2011 Sep;26(5):657-63. doi: 10.1007/s10103-011-0938-6. Epub 2011 May 31. PMID 21626017
- [Background] Youssef M, Ashkar S, Hamade E, Gutknecht N, Lampert F, Mir M. The effect of low-level laser therapy during orthodontic movement: a preliminary study. Lasers Med Sci. 2008 Jan;23(1):27-33. doi: 10.1007/s10103-007-0449-7. Epub 2007 Mar 15. PMID 17361391
- [Background] Sousa MV, Scanavini MA, Sannomiya EK, Velasco LG, Angelieri F. Influence of low-level laser on the speed of orthodontic movement. Photomed Laser Surg. 2011 Mar;29(3):191-6. doi: 10.1089/pho.2009.2652. Epub 2011 Jan 23. PMID 21254890
- [Background] Heravi F, Moradi A, Ahrari F. The effect of low level laser therapy on the rate of tooth movement and pain perception during canine retraction. Oral Health Dent Manag. 2014 Jun;13(2):183-8. PMID 24984620
- [Background] Whelan HT, Smits RL Jr, Buchman EV, Whelan NT, Turner SG, Margolis DA, Cevenini V, Stinson H, Ignatius R, Martin T, Cwiklinski J, Philippi AF, Graf WR, Hodgson B, Gould L, Kane M, Chen G, Caviness J. Effect of NASA light-emitting diode irradiation on wound healing. J Clin Laser Med Surg. 2001 Dec;19(6):305-14. doi: 10.1089/104454701753342758. PMID 11776448
- [Background] Weber JB, Pinheiro AL, de Oliveira MG, Oliveira FA, Ramalho LM. Laser therapy improves healing of bone defects submitted to autologous bone graft. Photomed Laser Surg. 2006 Feb;24(1):38-44. doi: 10.1089/pho.2006.24.38. PMID 16503787
- [Background] Saito S, Shimizu N. Stimulatory effects of low-power laser irradiation on bone regeneration in midpalatal suture during expansion in the rat. Am J Orthod Dentofacial Orthop. 1997 May;111(5):525-32. doi: 10.1016/s0889-5406(97)70152-5. PMID 9155812
- [Background] Masha RT, Houreld NN, Abrahamse H. Low-intensity laser irradiation at 660 nm stimulates transcription of genes involved in the electron transport chain. Photomed Laser Surg. 2013 Feb;31(2):47-53. doi: 10.1089/pho.2012.3369. Epub 2012 Dec 16. PMID 23240874
- [Background] Oron U, Ilic S, De Taboada L, Streeter J. Ga-As (808 nm) laser irradiation enhances ATP production in human neuronal cells in culture. Photomed Laser Surg. 2007 Jun;25(3):180-2. doi: 10.1089/pho.2007.2064. PMID 17603858
- [Background] Sun X, Zhu X, Xu C, Ye N, Zhu H. [Effects of low energy laser on tooth movement and remodeling of alveolar bone in rabbits]. Hua Xi Kou Qiang Yi Xue Za Zhi. 2001 Oct;19(5):290-3. Chinese. PMID 12539482

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OrthoPulse™ | Sham-Control OrthoPulse™
Started | 15 | 14
Completed | 14 | 12
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OrthoPulse™ | Sham-Control OrthoPulse™ | Total
Number analyzed (Participants) | 15 | 14 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.4 (1.5) | 13.3 (1.0) | 13.3 (1.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 7 | 5 | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 14 | 29

OUTCOME MEASURES:

1. Primary Outcome: Overall Orthodontic Treatment Time for OrthoPulse™ and Non-OrthoPulse™ Treated Patients.
Description: The amount of time that spans between the start of a patient's orthodontic treatment to when the qualified investigator deems the case complete, in that malocclusion is completely resolved and an acceptable clinical outcome is achieved.
Time Frame: Participants will be followed for the duration of their orthodontic treatment, an expected average of 1-2 years, depending on the severity of the case.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | OrthoPulse™ | Sham-Control OrthoPulse™
Number analyzed (Participants) | 14 | 12
months | 19.0 (5.5) | 21.2 (6.9)

ADVERSE EVENTS:
Time Frame: Whole study duration, 2 years.
Arm/Group | OrthoPulse™ | Sham-Control OrthoPulse™
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 0/15 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No